CLINICAL TRIAL: NCT02402699
Title: Ipilimumab 60-month Pharmacovigilance Protocol for Advanced Melanoma Patients Who Are Hepatitis B and/or Hepatitis C Virus Positive in Taiwan
Acronym: Yervoy RMP
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-414
Record Dates: First submitted 2015-03-16; First posted 2015-03-30 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Advanced Melanoma; Hepatitis B; Hepatitis C
Keywords: HBV; HBC
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unresectable, recurrent or metastatic melanoma patients: All adult unresectable, recurrent, or metastatic melanoma patients with HBV or HCV treated with at least 1 dose of ipilimumab therapy in Taiwan

SUMMARY:
This protocol is being conducted to comply with the direct request from the Taiwan Food and Drug Administration (TFDA) for a 60-month intensive pharmacovigilance protocol of patients with known hepatitis B (HBV) or hepatitis C (HCV) infection, regardless of control on antiviral therapy in Taiwan and who are treated with ipilimumab for advanced (unresectable, recurrent or metastatic) Melanoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Age of 18 years or older on date of first dose of Ipilimumab
* Patients who received at least 1 dose of Ipilimumab for the treatment of unresectable, recurrent or Metastatic Melanoma in Taiwan
* Patients with advanced Melanoma and HBV or HCV who are initiating Ipilimumab under the discretion of their physician

Exclusion Criteria:

* Patients who received Ipilimumab as part of a clinical trial
* Patients who are receiving Ipilimumab for any indication other than local approval (ie, unresectable or Metastatic Melanoma)
* Patients who are not infected with HBV or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult unresectable, recurrent, or Metastatic Melanoma patients with HBV or HCV treated with at least 1 dose of Ipilimumab therapy in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Identify and describe observed adverse events (AEs) based on liver function abnormalities and changes in hepatitis viral load | During 6months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Taipei, Taiwan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm